CLINICAL TRIAL: NCT02794506
Title: Propolis Improves Periodontal Status and Glycemic Control in Subjects With Type 2 Diabetes Mellitus and Chronic Periodontitis: a Randomized Clinical Trial
Brief Title: Propolis Improves Glycemic Control in Subjects With Type 2 Diabetes and Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Anees (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Anees, Lecturer of Oral Medicine and Periodontology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DENT-1971
Record Dates: First submitted 2016-05-29; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus; Periodontitis
Keywords: Diabetes mellitus; Chronic periodontitis; Propolis
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis; Chronic Periodontitis | interventions — Propolis; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propolis (Experimental): 400 mg oral proplois (capsule) was given to participants once daily for 6 months after performing scaling and root planing.
  Interventions: Drug: Propolis
- Placebo (Placebo Comparator): Placebo capsule was given to participants once daily for 6 months after performing scaling and root planing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propolis — Propolis capsules was taken by the experimental group for 6 months after receiving scaling and root planing (SRP).
  Other Names: BioPropolis
  Arms: Propolis
Drug: Placebo — Placebo capsules was taken by the control group for 6 months after receiving scaling and root planing (SRP).
  Other Names: Starch capsules
  Arms: Placebo

SUMMARY:
Background:

Propolis is a natural resin made by bees from various plant sources. Propolis exerts antimicrobial, anti-inflammatory, immunomodulatory, antioxidant, and antidiabetic properties. The purpose of this study was to assess the adjunctive benefit of propolis supplementation in individuals with both chronic periodontitis and type 2 diabetes mellitus (T2DM) receiving scaling and root planing (SRP).

Methods:

A 6-month randomized blinded clinical trial comparing SRP with placebo (placebo+SRP group, n=26) or combined with a 6- month regimen of 400 mg oral propolis once daily (propolis+SRP group, n=26) was performed in patients with long-standing T2DM and chronic periodontitis. Treatment outcomes included hemoglobin A1c (HbA1c), fasting plasma glucose (FPG), serum N€-(carboxymethyl) lysine (CML) and changes in periodontal parameters.

DETAILED DESCRIPTION:
INTRODUCTION

Diabetes mellitus (DM) is a metabolic disorder characterized by frequent periods of hyperglycemia, which induce certain molecular pathways that seem to be crucial to the initiation of angiopathic complications of DM. Several mechanisms have been suggested to explain the pathogenicity of complications of hyperglycemia such as protein kinase C isoforms, enhanced polyol pathway flux, and increased accumulation of advanced glycosylated end-products. A dysregulated immune response stemming from an inappropriate cytokine production is a possible mechanism underpinning the cross-susceptibility between periodontal disease and DM. DM has been unambiguously determined as one of the major risk factors of periodontitis. It was reported that the risk of periodontitis increases to almost threefold in diabetic patients when compared to healthy individuals. The glycemic control level is believed to be of paramount importance as a determinant of the increased risk for developing complications. Diabetic patients with an HbA1c level more than 9% were found to have an increased prevalence of advanced chronic periodontitis in comparison to healthy people according to the US National Health and Nutrition Examination Survey (NHANES) III.

Two decades ago, periodontitis was added to represent the sixth complication of DM. Individuals suffering from periodontal diseases often have increased serum levels of proinflammatory cytokines, such as IL-1, IL-6 and TNF-α. Diabetic patients with periodontitis possess hyperinflammatory immune cells that lead to enhanced release of proinflammatory cytokines, which eventually lead to insulin resistance resulting in a greater risk of poor glycemic control when compared to diabetic patients without periodontitis. The accumulation of irreversible advanced glycation end-products (AGEs), predominantly N€-(carboxymethyl) lysine (CML) has shown to alter cell function and tissue structure. Due to difficulty in managing diabetes; there is a critical need for new therapeutic modalities for prevention of diabetes-related complications.

Propolis is a natural resin synthesized by honey bees from substances extracted from parts of some plants, buds and sap. Due to its physical characteristics, propolis is utilized by the honey bees to protect the hives against foreign invaders. Propolis has been used for centuries as a homeopathic medicine known for its anti-inflammatory properties, especially in Europe and ancient Egypt. It has traditionally been used for the management of numerous diseases, such as gastrointestinal disorders and mucocutaneous infections of fungal, bacterial and viral etiology.

There are several types of propolis that differ in composition depending on the plant source which varies according to the geographic zone such as Brazil, Peru, China and Europe. Propolis contains more than more than 230 constituents, including flavonoids, cinnamic acids and their esters, caffeic acid and caffeic acid phenethyl ester. It has been found to have a wide array of biological activities, including antibacterial, antiviral, fungicidal, anti-inflammatory, antioxidant, hepatoprotective, free radical scavenging, immunomodulatory and anti-diabetic activity. Recently, investigations revealed that caffeic acid phenethyl ester (CAPE) is an important active molecule found in propolis and is responsible for most of its therapeutic properties.

The actions of Chinese and Brazilian propolis in streptozotocin-induced type 1 diabetes mellitus in Sprague Dawley rats was explored and the results indicated that both types of propolis significantly inhibited more body weight loss and plasma glucose increase in experimental rats. Additionally, rats treated with Chinese propolis exhibited an 8.4% reduction in HbA1c levels in comparison to non-treated diabetic group.

Hence, it was hypothesized that periodontal therapy with SRP in conjunction with oral daily supplementation of propolis in patients with chronic periodontitis and T2DM might improve both diabetic and periodontal outcomes. Thus, the aim of the current study is to evaluate whether the adjunctive therapy of oral propolis supplementation to SRP compared to SRP plus placebo, reduces glycated hemoglobin and improves clinical and periodontal parameters after 6 months of therapy in individuals with chronic periodontitis and T2DM.

MATERIALS AND METHODS

Study Population:

The study was approved by the Institutional Review Board of Mansoura University. Subjects were selected during their recall maintenance visits in the Internal Medicine Hospital, Mansoura University, between June and December in 2014. Patients filled out questionnaires gathering information on their dental and oral health care followed by a periodontal screening examination to determine eligible individuals. Patients were considered eligible for the study if they had T2DM with a minimum of five years duration and had been taking stable doses of oral hypoglycemic drugs and/or insulin for at least 6 months. In addition, they should have chronic periodontitis with probing pocket depth and clinical attachment loss ≥ 5 mm with detectable bleeding on probing in at least one site in each sextant. Patients should have a minimum of 20 teeth to be selected. All patients were diagnosed to have moderate to severe chronic periodontitis according to Armitage criteria (24). Exclusion criteria included smokers, recent extended use of antibiotics or non-steroidal anti-inflammatory drugs within the last 3 months, patients who had any periodontal therapy within one year, patients with grade 3 or 4 retinopathy, pregnancy or women using oral contraceptives. Enrolled patients signed written informed consents for study participation.

Study Design:

Fifty two people with T2DM diagnosed with moderate to severe chronic periodontitis were randomly assigned using computer-generated random tables to receive propolis (400 mg capsule orally once daily for six months) as adjuvant to scaling and root planing (Propolis+ SRP group, n = 26), or matching placebo capsules for 6 months in addition to scaling and root planing (Placebo+SRP group, n = 26) in this parallel randomized blinded controlled trial with an allocation ratio = 1:1. The generated allocation sequences were concealed in closed stapled envelopes until interventions were assigned. Investigators were not involved during randomization. Propolis commercially named BioPropolis (Sigma Pharmaceutical Industries for International Business Establishment Co. IBE Pharma, Cairo, Egypt) and matching placebo capsules were used in the study. All participants in both groups were assigned to receive equal number of capsules during the 6- month period. Vials which contain propolis and placebo drugs were labeled with specific codes unknown to patients and investigators. Patients were instructed to take only one capsule daily from the given vial. Patient compliance was calculated by counting the remaining capsules in each returned vial every month. Untoward side effects of both medications were queried and recorded at each visit during the study period.

All individuals received meticulous full mouth scaling and root planing (SRP) with hand curettes and ultrasonic tips under local anesthesia until root surfaces were smooth by clinician (MA) in a single visit. Oral hygiene instructions and motivations for proper tooth brushing and dental flossing were given to the patients. Chlohexidine 0.12% mouthrinse was prescribed for all patients for only two weeks after SRP.

Clinical Periodontal Measurements:

Clinical periodontal parameters including probing pocket depth (PD), clinical attachment level (CAL) (distance from the CEJ to the base of the pocket), Eastman interdental bleeding (EIBI) , gingival (GI) and plaque (PI) indices were assessed at baseline, 3 months and 6 months after therapy by the examiner (HE). Intra-examiner calibration was achieved by examination of 10 patients twice, 24 hours apart before starting the study. Calibration was accepted if measurements of PD and CAL (by using UNC-15 probe) at baseline and 24 hours were similar to 1 mm at the 90% level.

Collection and analysis of Blood:

10 mL of venous blood from the antecubital vein of all participants were collected in heparinized vacutainer tubes at baseline, 3 months and 6 months after treatment. Measurements of HbA1c were carried out via an automated affinity chromatography system (Bio-Rad Micromat II, Hercules, CA). Fasting plasma glucose levels (FPG) were measured by the standard glucose oxidase method. The serum concentration of N€-(carboxymethyl) lysine (CML) was assessed by N€-(carboxymethyl) lysine (CML) ELISA Kit of CML protein adducts (OxiSelect™, Catalog Number STA-316, Cell Biolabs Inc., San Diego, CA, USA). The amount of CML adduct in protein samples was evaluated by comparing the absorbance to a known CML-BSA standard curve as described by the manufacturer.

Study outcomes:

The primary outcome of the present clinical trial was the change in HbA1c levels after 6 months of therapy. Secondary outcomes included the change in HbA1c levels after 3 months in addition to the amount of CAL gain, PD reduction and changes in FPG and serum CML levels after 3 and 6 months of therapy.

Statistical Analysis:

A power analysis was performed before commencement of the trial with type I error α = 0.05, β = 0.14 and (1-β) = 0.86. The power was calculated as p = 0.8641 and the estimated minimum sample size required was found to be 20 per each group to achieve a power of 80% based on achievement of 6-month reduction of HbA1c of the test group over the control by 0.8%. All data were explored by using Kolmogrov-Smirnov test of normality. Parametric data were presented as mean ± SD. Baseline comparisons were made using Student's t-test. One-way analyses of variance (ANOVA) with Holm-Sidak post hoc correction for multiple comparisons were used to determine significant changes at different time intervals. Wilcoxon signed rank test and Mann-Whitney test were used to detect differences per group and between groups over time. The α-level for significance was set at 0.05.Statistical analyses were calculated by a statistical software program (Statistical Package for the Social Sciences version 19.0, SPSS, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Patients had type 2 diabetes mellitus with a minimum of five years duration and had been taking stable doses of oral hypoglycemic drugs and/or insulin for at least 6 months.
* Patients should have chronic periodontitis with probing pocket depth and clinical attachment loss ≥ 5 mm with detectable bleeding on probing in at least one site in each sextant.
* Patients should have a minimum of 20 teeth to be selected.
* All patients were diagnosed to have moderate to severe chronic periodontitis according to Armitage criteria.

Exclusion Criteria:

* Smokers.
* Recent extended use of antibiotics or non-steroidal anti-inflammatory drugs within the last 3 months.
* Patients who had any periodontal therapy within one year.
* Patients with grade 3 or 4 retinopathy.
* Pregnancy.
* Women using oral contraceptives.

Ages: 38 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of glycosylated hemoglobin (HbA1c) | Baseline, 3 and 6 months
  HbA1c was evaluated at baseline,3 and 6 months

SECONDARY OUTCOMES:
Change of pocket depth | From baseline and 6 months
Change of clinical attachment level | From baseline and 6 months
Change of fasting plasma glucose level | From baseline and 6 months
Change of serum N- epsilon (carboxymethyl) lysine level | From baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M. El-Sharkawy, Ass.Prof., Study Director — Mansoura University
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Schalkwijk CG, Stehouwer CD. Vascular complications in diabetes mellitus: the role of endothelial dysfunction. Clin Sci (Lond). 2005 Aug;109(2):143-59. doi: 10.1042/CS20050025. PMID 16033329
- [Background] Piarulli F, Sartore G, Lapolla A. Glyco-oxidation and cardiovascular complications in type 2 diabetes: a clinical update. Acta Diabetol. 2013 Apr;50(2):101-10. doi: 10.1007/s00592-012-0412-3. Epub 2012 Jul 5. PMID 22763581
- [Background] Folli F, Corradi D, Fanti P, Davalli A, Paez A, Giaccari A, Perego C, Muscogiuri G. The role of oxidative stress in the pathogenesis of type 2 diabetes mellitus micro- and macrovascular complications: avenues for a mechanistic-based therapeutic approach. Curr Diabetes Rev. 2011 Sep;7(5):313-24. doi: 10.2174/157339911797415585. PMID 21838680
- [Background] Hegab Z, Gibbons S, Neyses L, Mamas MA. Role of advanced glycation end products in cardiovascular disease. World J Cardiol. 2012 Apr 26;4(4):90-102. doi: 10.4330/wjc.v4.i4.90. PMID 22558488
- [Background] Mahanonda R, Pichyangkul S. Toll-like receptors and their role in periodontal health and disease. Periodontol 2000. 2007;43:41-55. doi: 10.1111/j.1600-0757.2006.00179.x. No abstract available. PMID 17214834
- [Background] Soskolne WA, Klinger A. The relationship between periodontal diseases and diabetes: an overview. Ann Periodontol. 2001 Dec;6(1):91-8. doi: 10.1902/annals.2001.6.1.91. PMID 11887477
- [Background] Salvi GE, Yalda B, Collins JG, Jones BH, Smith FW, Arnold RR, Offenbacher S. Inflammatory mediator response as a potential risk marker for periodontal diseases in insulin-dependent diabetes mellitus patients. J Periodontol. 1997 Feb;68(2):127-35. doi: 10.1902/jop.1997.68.2.127. PMID 9058329
- [Background] Negishi J, Kawanami M, Terada Y, Matsuhashi C, Ogami E, Iwasaka K, Hongo T. Effect of lifestyle on periodontal disease status in diabetic patients. J Int Acad Periodontol. 2004 Oct;6(4):120-4. PMID 15553978
- [Background] Garcia D, Tarima S, Okunseri C. Periodontitis and glycemic control in diabetes: NHANES 2009 to 2012. J Periodontol. 2015 Apr;86(4):499-506. doi: 10.1902/jop.2014.140364. Epub 2014 Nov 27. PMID 25427615
- [Background] Loe H. Periodontal disease. The sixth complication of diabetes mellitus. Diabetes Care. 1993 Jan;16(1):329-34. No abstract available. PMID 8422804
- [Background] Chen L, Chen R, Wang H, Liang F. Mechanisms Linking Inflammation to Insulin Resistance. Int J Endocrinol. 2015;2015:508409. doi: 10.1155/2015/508409. Epub 2015 Jun 2. PMID 26136779
- [Background] Mendez JD, Xie J, Aguilar-Hernandez M, Mendez-Valenzuela V. Trends in advanced glycation end products research in diabetes mellitus and its complications. Mol Cell Biochem. 2010 Aug;341(1-2):33-41. doi: 10.1007/s11010-010-0434-5. Epub 2010 Mar 23. PMID 20309613
- [Background] Miao M, Niu Y, Xie T, Yuan B, Qing C, Lu S. Diabetes-impaired wound healing and altered macrophage activation: a possible pathophysiologic correlation. Wound Repair Regen. 2012 Mar-Apr;20(2):203-13. doi: 10.1111/j.1524-475X.2012.00772.x. PMID 22380690
- [Background] Gabrys J, Konecki J, Krol W, Scheller S, Shani J. Free amino acids in bee hive product (propolis) as identified and quantified by gas-liquid chromatography. Pharmacol Res Commun. 1986 Jun;18(6):513-8. doi: 10.1016/0031-6989(86)90146-3. PMID 3749241
- [Background] Sanghani NN, Bm S, S S. Health from the hive: propolis as an adjuvant in the treatment of chronic periodontitis - a clinicomicrobiologic study. J Clin Diagn Res. 2014 Sep;8(9):ZC41-4. doi: 10.7860/JCDR/2014/8817.4856. Epub 2014 Sep 20. PMID 25386520
- [Background] Santos VR, Pimenta FJ, Aguiar MC, do Carmo MA, Naves MD, Mesquita RA. Oral candidiasis treatment with Brazilian ethanol propolis extract. Phytother Res. 2005 Jul;19(7):652-4. doi: 10.1002/ptr.1715. PMID 16161031
- [Background] Coelho LG, Bastos EM, Resende CC, Paula e Silva CM, Sanches BS, de Castro FJ, Moretzsohn LD, Vieira WL, Trindade OR. Brazilian green propolis on Helicobacter pylori infection. a pilot clinical study. Helicobacter. 2007 Oct;12(5):572-4. doi: 10.1111/j.1523-5378.2007.00525.x. PMID 17760728
- [Background] Nolkemper S, Reichling J, Sensch KH, Schnitzler P. Mechanism of herpes simplex virus type 2 suppression by propolis extracts. Phytomedicine. 2010 Feb;17(2):132-8. doi: 10.1016/j.phymed.2009.07.006. Epub 2009 Aug 13. PMID 19682876
- [Background] Banskota AH, Tezuka Y, Adnyana IK, Midorikawa K, Matsushige K, Message D, Huertas AA, Kadota S. Cytotoxic, hepatoprotective and free radical scavenging effects of propolis from Brazil, Peru, the Netherlands and China. J Ethnopharmacol. 2000 Sep;72(1-2):239-46. doi: 10.1016/s0378-8741(00)00252-x. PMID 10967477
- [Background] Czyzewska U, Kononczuk J, Teul J, Dragowski P, Pawlak-Morka R, Surazynski A, Miltyk W. Verification of chemical composition of commercially available propolis extracts by gas chromatography-mass spectrometry analysis. J Med Food. 2015 May;18(5):584-91. doi: 10.1089/jmf.2014.0069. Epub 2014 Sep 8. PMID 25198412
- [Background] Zhu W, Chen M, Shou Q, Li Y, Hu F. Biological activities of chinese propolis and brazilian propolis on streptozotocin-induced type 1 diabetes mellitus in rats. Evid Based Complement Alternat Med. 2011;2011:468529. doi: 10.1093/ecam/neq025. Epub 2011 Apr 14. PMID 21785625
- [Background] Armutcu F, Akyol S, Ustunsoy S, Turan FF. Therapeutic potential of caffeic acid phenethyl ester and its anti-inflammatory and immunomodulatory effects (Review). Exp Ther Med. 2015 May;9(5):1582-1588. doi: 10.3892/etm.2015.2346. Epub 2015 Mar 11. PMID 26136862
- [Background] Tolba MF, Azab SS, Khalifa AE, Abdel-Rahman SZ, Abdel-Naim AB. Caffeic acid phenethyl ester, a promising component of propolis with a plethora of biological activities: a review on its anti-inflammatory, neuroprotective, hepatoprotective, and cardioprotective effects. IUBMB Life. 2013 Aug;65(8):699-709. doi: 10.1002/iub.1189. Epub 2013 Jul 11. PMID 23847089
- [Background] Armitage GC. Periodontal diagnoses and classification of periodontal diseases. Periodontol 2000. 2004;34:9-21. doi: 10.1046/j.0906-6713.2002.003421.x. No abstract available. PMID 14717852
- [Background] Abrams K, Caton J, Polson A. Histologic comparisons of interproximal gingival tissues related to the presence or absence of bleeding. J Periodontol. 1984 Nov;55(11):629-32. doi: 10.1902/jop.1984.55.11.629. PMID 6334156
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Rosevear JW, Pfaff KJ, Service FJ, Molnar GD, Ackerman E. Glucose oxidase method for continuous automated blood glucose determination. Clin Chem. 1969 Aug;15(8):680-98. No abstract available. PMID 5808451